CLINICAL TRIAL: NCT02362100
Title: Proximal Humerus Fractures Randomized Control Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to low recruitment, lack of funding, and challenges maintaining follow-up in this patient population, a decision was made to terminate this study.
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20150458-01H
Record Dates: First submitted 2015-02-08; First posted 2015-02-12 (Estimated); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Proximal Humerus Fracture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nonoperative management (Placebo Comparator): Treatment will consist of sling immobilization for a period of 6 weeks. Details and treatment timeline as follows:
  * 0 - 3 weeks: immobilization with a shoulder sling, range of motion of elbow, hand and wrist
  * 3 - 6 weeks: same as 0-3 weeks, with addition of pendulum exercises every two hours
  * After 6 weeks: Active mobilization and removal of sling. Light activity permitted and physiotherapy for range of motion permitted as tolerated.
  * After 6 months: no further restriction will be placed. Full home and work activity permitted.
  Interventions: Other: Non operative
- locking plate surgical fixation (Active Comparator): Standardized operative management protocol as follows:
  * Pre-operative medical clearance established via anesthesia consults if required for medically complex patients.
  * Provision of pre-operative intravenous (IV) antibiotic prophylaxis:
  * Administration of general anesthetic.
  * Patient positioning and preparation:
    * Patient is carefully placed in the beach-chair position,
    * Deltopectoral approach Fracture reduction and fixation with confirmation with intraoperative fluoroscopy images.
  Interventions: Procedure: locking plate surgical fixation

INTERVENTIONS:
Other: Non operative — non operative treatment
  Arms: nonoperative management
Procedure: locking plate surgical fixation
  Arms: locking plate surgical fixation

SUMMARY:
The primary objective is to determine if a difference exists in functional outcomes, as measured by the Constant score, when comparing nonoperative management and locking plate surgical fixation of low-energy displaced proximal humerus fractures in the elderly population over a 2-year follow-up period. Secondary outcomes will include an assessment of the ASES score, the SF-36 quality of life score, complication rates, re-operation rates, radiographic time to union, radiographic malunion, hardware position and evidence of avascular necrosis or posttraumatic osteoarthritis .

DETAILED DESCRIPTION:
The design of this study is two-fold. The main study will be a prospective, single blind, randomized controlled trial (RCT). Patients will be randomized to either (1) non-operative treatment or (2) locking plate open reduction and internal fixation (ORIF).

The second component of this study will be a prospective, cohort study. This option will be presented to patients who do not want to enroll in the RCT because they prefer one treatment option over the other, and do not wish to be randomized to a treatment. Patients who choose either non-operative treatment or ORIF for their proximal humerus fracture will be followed for 2 years post injury.

Study Objectives:

Objective 1: Does a difference exist in the functional outcome between non-operative management and locking plate surgical fixation of low-energy displaced two-part, three-part, and four-part proximal humerus fractures in the elderly population based on the Constant functional outcome score over a 2-year follow-up period? Objective 2: Does a difference exist between non-operative management and locking plate surgical fixation of low-energy displaced two-part, three-part, and four-part proximal humerus fractures in the elderly population based on the ASES functional outcome score, the short form Patient Reported Outcomes Measurement Information System (PROMIS) upper extremity score, the International Physical Activity Questionnaire (IPAQ) for the elderly, and the EuroQol EQ-5D-5L Health Questionnaire Quality of Life (QoL) functional outcome score over a 2-year follow-up period? What is the incidence of complications of non-operative management and locking plate surgical fixation of low-energy displaced two-part, three-part, and four-part proximal humerus fractures in the elderly population based on infection, nerve injury, intra-articular screw penetration and bleeding (hematoma), reoperation rate, or hospital readmission over a 2-year follow-up period? Objective 3: Does a difference exist between non-operative management and locking plate surgical fixation of low-energy displaced two-part, three-part, and four-part proximal humerus fractures in the elderly population based on radiographic outcomes including non-union, malunion, and joint arthrosis? Objective 4: Does the degree of initial displacement or angulation of the fracture fragments correlate with final functional outcome measures? Objective 5: Does the quality of the surgical reduction correlate with final functional outcome measures?

ELIGIBILITY:
Inclusion Criteria:

1. Displaced 2- or 3-part proximal humerus fractures by the Neer classification.
2. Displaced 4-part proximal humeral fractures by the Neer classification that are deemed amenable to surgical fixation.
3. > 60 years of age
4. Low energy mechanism of injury
5. Acute fracture (<3 weeks)

Exclusion Criteria:

1. 4-part proximal humerus fractures that are not deemed amenable to surgical fixation (eg. due to osteopenic bone, thin head or tuberosity fragments); fractures that are better suited to treatment with arthroplasty
2. Isolated greater tuberosity fractures
3. Ipsilateral upper extremity significant injury, concomitant fracture or polytrauma
4. Open fracture
5. Previous ipsilateral shoulder surgery
6. Patients with active worker's compensation claims (due to the expectation of lower rates of success in this patient population)
7. Active joint or systemic infection
8. Patients with convulsive disorders, collagen diseases, and any other conditions that might affect the mobility of the shoulder joint
9. Major medical illness (life expectancy less than 2 years, unacceptably high operative risk, or not medically cleared by preoperative anesthesia consult)
10. Unable to speak or read English/French
11. Psychiatric illness that precludes informed consent
12. Unwilling to be followed for 2 years

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Change in Constant Score | From baseline to up until 24-Months Post-Operative
  The Constant Score reflects an overall clinical functional assessment. This instrument is based on a 100-point scoring system. Subjective findings (pain, activities of daily living, and working in different positions) make up a total of 35 points. Objective measurements make up the remaining 65 points.The test is divided into four sub-categories: (1) pain is measured using 4 likert levels (15 points maximum), where a higher score indicates a better outcome; activities of daily living are measured using a likert scale, where a higher number indicates better outcomes (20 points maximum); mobility is measured by an assessor, and rated using a likert scale where a higher score indicates better outcomes (40 points maximum); finally, strength is measured by an assessor where 1 point is given per 0.5kg of force (maximum 25 points), a higher score indicates better outcomes. All categories are added together, and a total score out of 100 is given (higher score indicates better outcome).

SECONDARY OUTCOMES:
Change in American Shoulder and Elbow Surgeons Standardized Shoulder Assessment | From baseline to up until 24-Months Post-Operative
  The ASES is a shoulder specific assessment divided into two sections: pain and activities of daily living (ADL). Pain is recorded on a visual analogue scale (0-10), lower scores indicate better outcomes. There are 10 activities of daily living questions, each are recorded on a 4 level likert scale (0-3), which a higher score indicates a better outcome. The overall score is an equal weight of the two sections and produces a score out of 100. The higher the score, the better the outcome.
Change in Short Form-36 | From baseline to up until 24-Months Post-Operative
  The Short Form 36 (SF-36) is an outcome measure used to determine quality of life. This measure has 8 scaled scores, each question has equal weight and is then translated onto a scale graded from 0-100. A higher number indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lapner, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196
- [Derived] Howard L, Berdusco R, Momoli F, Pollock J, Liew A, Papp S, Lalonde KA, Gofton W, Ruggiero S, Lapner P. Open reduction internal fixation vs non-operative management in proximal humerus fractures: a prospective, randomized controlled trial protocol. BMC Musculoskelet Disord. 2018 Aug 18;19(1):299. doi: 10.1186/s12891-018-2223-3. PMID 30121091